CLINICAL TRIAL: NCT04234672
Title: A Phase 1 Study to Assess Absolute Bioavailability of TAK-831 and to Characterize Mass Balance, Pharmacokinetics, Metabolism, and Excretion of [14C]TAK-831 in Male Healthy Subjects
Brief Title: A Study to Assess Absolute Bioavailability (ABA) of TAK-831 and to Characterize Mass Balance, Pharmacokinetics (PK), Metabolism, and Excretion of [14C]TAK-831 in Male Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Neurocrine Biosciences (Industry)
Collaborators: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: TAK-831-1008; U1111-1242-9877 (Registry Identifier: WHO)
Record Dates: First submitted 2020-01-16; First posted 2020-01-21 (Actual); Results first posted 2021-04-28 (Actual); Last update posted 2021-06-30 (Actual); Status verified 2021-06

CONDITIONS: Healthy Volunteers
Keywords: Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg (Experimental): TAK-831 500 mg, tablet, orally, once on Day 1, followed by [14C]TAK-831 50 micrograms (μg) [approximately 1 microcurie (μCi)], infusion, intravenously (IV), once on Day 1 of Treatment Period 1, followed by a washout period of 8 days, further followed by [14C]TAK-831 500 mg (approximately 100 μCi), suspension, orally, once under fasted state on Day 1 of Treatment Period 2.
  Interventions: Drug: TAK-831 Oral Tablet; Drug: [14C]TAK-831 IV Infusion; Drug: [14C]TAK-831 Oral Suspension

INTERVENTIONS:
Drug: TAK-831 Oral Tablet — TAK-831 tablet.
  Other Names: Luvadaxistat
Drug: [14C]TAK-831 IV Infusion — [14C]TAK-831 IV infusion.
Drug: [14C]TAK-831 Oral Suspension — [14C]TAK-831 oral suspension.

SUMMARY:
The purpose of this study is to determine ABA of TAK-831 following a single microdose intravenous administration of 50 microgram (μg) (approximately 1 microcurie [μCi]) [14C]TAK-831 and a single oral administration of 500 milligram (mg) TAK-831 tablets in Period 1, and to assess the mass balance, characterize the PK of TAK-831 in plasma and urine, and total radioactivity concentration equivalents in plasma and whole blood following a single oral suspension dose of 500 mg (approximately 100 μCi) [14C]TAK-831 in Period 2.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-831 (also known as luvadaxistat). The study will determine ABA in Period 1, and the absorption, metabolism, excretion, and mass balance of TAK-831 after single oral administration in Period 2 in healthy adult male participants, by collecting plasma, urine, and feces samples for drug concentration analysis, and plasma, whole blood, urine, and fecal samples for total radioactivity analysis and metabolic profiling.

The study will enroll approximately 6 participants. The study is designed to consist of 2 periods: Period 1 (ABA study period) and Period 2 (absorption, distribution, metabolism, and elimination [ADME] study period). In Period 1 (ABA study period), all participants will receive a single unlabelled oral dose of TAK-831 as tablet and a microdose intravenous infusion of 50 μg (approximately 1 μCi) [14C]TAK-831, followed by a washout period of 8 days before the dose in Period 2. In Period 2 (ADME study period), all participants will receive a single dose of 500 mg (approximately 100 μCi) [14C]TAK-831 as an oral suspension.

This single center trial will be conducted in the United States. The overall time to participate in this study is approximately 65 days including screening period. Participants will be contacted approximately 30 days after the last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

1. Weighs at least 45 kilogram (kg) and body mass index (BMI) greater than or equal to (>=) 18.0 and less than (˂) 32.0 kilogram per square meter (kg/m^2) at screening.

Exclusion Criteria:

1. Seated blood pressure is less than 90/40 millimeter of mercury (mmHg) or greater than 140/90 mmHg at screening.
2. Seated heart rate is lower than 40 beats per minute (bpm) or higher than 99 bpm at screening.
3. Estimated creatinine clearance <80 milliliter per minute (mL/min) at screening.
4. Has tattoo(s) or scarring at or near the site of intravenous infusion or any other condition which may interfere with infusion site examination, in the opinion of the Investigator.
5. Has infrequent bowel movements (less than approximately once per day) within 30 days prior to first dosing.
6. Has received radiolabeled substances or has been exposed to radiation sources within 12 months of first dosing or is likely to receive radiation exposure or radioisotopes within 12 months of first dosing such that participation in this study would increase their total exposure beyond the recommended levels considered safe (that is weighted annual limit recommended by the International Commission on Radiological Protection [ICRP] of 3000 milli roentgen equivalent man [mrem]).
7. Has been on a diet incompatible with the on-study diet, in the opinion of the Investigator or designee, within the 30 days prior to the first dosing and throughout the study.
8. Donation of blood or significant blood loss within 56 days prior to the first dosing.
9. Plasma donation within 7 days prior to the first dosing.

Ages: 19 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 6 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-04 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Celerion, Lincoln, Nebraska, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in the United States from 17 Feb 2020 to 04 April 2020.
Pre-assignment Details: Healthy male participants were enrolled in this study to receive TAK-831 tablets followed by radio-labelled TAK-831 intravenous (IV) infusion on Day 1 of Treatment Period 1 and radio-labelled TAK-831 oral suspension on Day 1 of Treatment Period 2. There was an 8-day washout period between the two periods.
Groups:
- TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg: TAK-831 5 X 100 mg tablets, orally, once on Day 1, followed by [14C]TAK-831 50 micrograms (μg) [approximately 1 microcurie (μCi)], infusion, intravenously (IV), once on Day 1 of Treatment Period 1, followed by a washout period of 8 days, further followed by [14C]TAK-831 500 mg (approximately 100 μCi), suspension, orally, once under fasted state on Day 1 of Treatment Period 2.
Period: Treatment Period 1 (Day 1)
Arm/Group | TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Washout Period (Day 2 to 8)
Arm/Group | TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg
Started | 6
Completed | 6
Not Completed | 0
Period: Treatment Period 2(Day9[Day1of Period2])
Arm/Group | TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety Population included all participants who received at least one dose of the study drug.
Arm/Group | TAK-831 500 mg + [14C]TAK-831 50 μg + [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.2 (6.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 3
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 6
Height [Mean (Standard Deviation); unit: cm] | 174.8 (6.1)
Weight [Mean (Standard Deviation); unit: kg] | 80.25 (6.5)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] — BMI = weight (kg)/[height (m)^2]
  kg/m^2 | 26.28 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Period 1: Percent Absolute Bioavailability (%F) for TAK-831
Description: Bioavailability is defined as the proportion of a drug which enters the circulation when introduced into the body and so is able to have an active effect. Percent absolute bioavailability, calculated for plasma TAK-831 as [Actual Dose (IV) x AUCinf (oral)] / [Actual Dose (oral) x AUCinf (IV)] x 100.
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours) post-dose in Treatment Period 1
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the oral dose of TAK-831 5 X 100 mg tablets and 50 ug IV dose in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percent absolute bioavailability
Groups:
- TAK-831 500 mg + [14C]TAK-831 50 μg: TAK-831 5 X 100 mg tablets, orally, followed by [14C]TAK-831 50 μg (approximately 1 μCi), 15-minute IV infusion, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-831 500 mg + [14C]TAK-831 50 μg
Number analyzed (Participants) | 6
percent absolute bioavailability | 17.34 (31.3)

2. Primary Outcome: Period 2: Total Radioactivity Expressed as Cumulative Percentage of Dose of [14C]TAK-831 Eliminated in Urine and Feces Combined [Combined Cum%Dose]
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the oral dose of [14C]TAK-831 500 mg oral suspension in Treatment Period 2 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Groups:
- [14C]TAK-831 500 mg: [14C]TAK-831 500 mg (approximately 100 μCi), suspension, orally, under fasted state, once on Day 1 of Treatment Period 2.
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
percentage of dose | 88.66 (3.6)

3. Primary Outcome: Period 2: Total Radioactivity Expressed as Cumulative Amount of [14C]TAK-831 Eliminated in Urine and Feces Combined (Combined CumAe)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg equivalents (eq) of parent drug
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
mg equivalents (eq) of parent drug | 472.7 (3.3)

4. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose of [14C]TAK-831 Excreted in Urine (Cum%Dose [UR])
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
percentage of dose | 27.50 (19.8)

5. Primary Outcome: Period 2: Percentage of Administered Radioactive Dose of [14C]TAK-831 Excreted in Feces (Cum%Dose [Fe])
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: percentage of dose
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
percentage of dose | 60.71 (5.9)

6. Primary Outcome: Period 2: Cmax: Maximum Observed Plasma Concentration of TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng/mL | 1243 (33.2)

7. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) of TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hours (hr)
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hours (hr) | 0.799 [0.52 to 1.05]

8. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of TAK-831 in Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 10.314 (6.3900)

9. Primary Outcome: Period 2: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity of TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng*hr/mL | 4198 (30.8)

10. Primary Outcome: Period 2: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration of TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng*hr/mL | 4171 (30.8)

11. Primary Outcome: Period 2: Cmax: Maximum Observed Plasma Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq/mL | 5878 (11.4)

12. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Plasma Radioactivity Concentration (Cmax)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 2.005 [1.01 to 4.17]

13. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Plasma Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 3.162 (0.3068)

14. Primary Outcome: Period 2: AUCinf: Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Infinity
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 31010 (9.8)

15. Primary Outcome: Period 2: AUClast: Area Under the Plasma Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/mL
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq*hr/mL | 28860 (8.8)

16. Primary Outcome: Period 2: Cmax: Maximum Observed Whole Blood Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq/g
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq/g | 2881 (9.2)

17. Primary Outcome: Period 2: Tmax: Time to Reach the Maximum Whole Blood Radioactivity Concentration (Cmax)
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Median (Full Range); unit: hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 2.001 [2.00 to 4.15]

18. Primary Outcome: Period 2: t(1/2)z: Terminal Disposition Phase Half-life of Whole Blood Radioactivity Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 2.580 (0.3922)

19. Primary Outcome: Period 2: AUCinf: Area Under the Whole Blood Radioactivity Concentration-time Curve From Time 0 to Infinity
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/g
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq*hr/g | 15180 (13.7)

20. Primary Outcome: Period 2: AUClast: Area Under the Whole Blood Radioactivity Concentration-time Curve From Time 0 to Last Quantifiable Concentration
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose in Treatment Period 2
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng eq*hr/g
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
ng eq*hr/g | 13420 (14.2)

21. Primary Outcome: Period 2: CLR: Renal Clearance for TAK-831 in Urine
Time Frame: Day 1 pre-dose and at multiple time points (up to 240 hours) post-dose
Population: as for outcome 2
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/hr
Arm/Group | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6
L/hr | 0.06547 (38.6)

22. Secondary Outcome: Period 1: Ceoi: Plasma Concentration at the End of Infusion for [14C]TAK-831
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the [14C]TAK-831 50 μg IV infusion in Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: picograms per milliliter (pg/mL)
Groups:
- [14C]TAK-831 50 μg: [14C]TAK-831 50 μg (approximately 1 μCi), infusion, 15-minute IV infusion, once on Day 1 of Treatment Period 1 after the TAK-831 oral dose, followed by a washout period of at least 7 days.
Arm/Group | [14C]TAK-831 50 μg
Number analyzed (Participants) | 6
picograms per milliliter (pg/mL) | 2903 (26.7)

23. Secondary Outcome: Period 1: Cmax: Maximum Observed Plasma Concentration for TAK-831 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours) post-dose in Treatment Period 1
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the oral dose of TAK-831 5 X 100 mg tablets in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Groups:
- TAK-831 500 mg: TAK-831 500 mg, tablet, orally, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-831 500 mg
Number analyzed (Participants) | 6
ng/mL | 1121 (45.5)

24. Secondary Outcome: Period 1: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for TAK-831 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours) post-dose in Treatment Period 1
Population: as for outcome 23
Measure: Median (Full Range); unit: hr
Arm/Group | TAK-831 500 mg
Number analyzed (Participants) | 6
hr | 1.255 [0.50 to 2.10]

25. Secondary Outcome: Period 1: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for TAK-831 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours) post-dose in Treatment Period 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanogram hour/milliliter (ng*hr/mL)
Arm/Group | TAK-831 500 mg
Number analyzed (Participants) | 6
nanogram hour/milliliter (ng*hr/mL) | 3436 (45.7)

26. Secondary Outcome: Period 1: AUCinf: Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for [14C]TAK-831 After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the [14C]TAK-831 50 ug IV dose in Treatment Period 1 were evaluated for this outcome measure.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | [14C]TAK-831 50 μg
Number analyzed (Participants) | 6
pg*hr/mL | 1992 (18.1)

27. Secondary Outcome: Period 1: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for TAK-831 After Oral Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours) post-dose in Treatment Period 1
Population: as for outcome 23
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*hr/mL
Arm/Group | TAK-831 500 mg
Number analyzed (Participants) | 6
ng*hr/mL | 3397 (46.6)

28. Secondary Outcome: Period 1: AUClast: Area Under the Plasma Concentration-time Curve From Time 0 to Last Quantifiable Concentration for [14C]TAK-831 After IV Administration
Time Frame: Day 1 pre-dose and at multiple time points (up to 95 hours) post-dose in Treatment Period 1
Population: as for outcome 26
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: pg*hr/mL
Arm/Group | [14C]TAK-831 50 μg
Number analyzed (Participants) | 6
pg*hr/mL | 1972 (18.1)

29. Secondary Outcome: Period 1: t(1/2)z: Terminal Disposition Half-life for TAK-831 After Oral and [14C]TAK-831 After IV Administration in Plasma
Time Frame: Day 1 pre-dose and at multiple time points (up to 96.5 hours for TAK-831 and up to 95 hours for [14C]TAK-831) post-dose
Population: PK-evaluable population included all participants who complied sufficiently with the protocol and displayed an evaluable PK profile. Participants who received the oral dose of TAK-831 5 X 100 mg tablets and [14C]TAK-831 50 ug IV dose in Treatment Period 1 were evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg
Number analyzed (Participants) | 6 | 6
hr | 12.278 (6.0291) | 3.815 (1.0456)

30. Secondary Outcome: Number of Participants Reporting One or More Treatment-emergent Adverse Events (TEAEs)
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE is defined as an AE with an onset that occurs after receiving study drug.
Time Frame: From first dose of study drug up to 30 days after last dose of study drug (up to approximately 38 days)
Population: Safety Population included all participants who received at least one dose of the study drug. Data is reported as per the treatment received in Treatment Periods 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 2

31. Secondary Outcome: Number of Participants With TEAEs Related to Electrocardiogram (ECG)
Description: The ECG parameters were considered TEAEs if they were judged to be clinically significant (i.e., if some action or intervention was required or if the Investigator judged the change to be beyond the range of normal physiologic fluctuation).
Time Frame: Up to Day 14
Population: Safety Population included all participants who received at least one dose of the study drug and will be included in the safety evaluations. Data is reported as per the treatment received in Treatment Periods 1 and 2.
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

32. Secondary Outcome: Number of Participants With TEAEs Related to Vital Signs
Description: Vital Signs included body temperature, respiratory rate, blood pressure, and heart rate. Any clinically significant changes from Baseline as assessed by the investigator were reported as TEAEs.
Time Frame: Up to Day 14
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

33. Secondary Outcome: Number of Participants With TEAEs Related to Laboratory Parameters
Description: The laboratory parameters included parameters of hematology, serum checmistry and urinalysis. The laboratory parameters were considered TEAEs if their values were judged to be clinically significant (i.e., if some action or intervention was required or if the Investigator judged the change to be beyond the range of normal).
Time Frame: Up to Day 14
Population: as for outcome 31
Measure: Count of Participants; unit: Participants
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg | [14C]TAK-831 500 mg
Number analyzed (Participants) | 6 | 6 | 6
Participants | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From first dose of study drug up to 30 days after last dose of the study drug (up to approximately 38 days)
Description: Data is reported as per the treatment received in Periods 1 and 2.
Groups:
- TAK-831 500 mg: TAK-831 5 X 100 mg tablets, orally, once on Day 1 of Treatment Period 1.
Arm/Group | TAK-831 500 mg | [14C]TAK-831 50 μg | [14C]TAK-831 500 mg
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TAK-831 500 mg (N=6) | [14C]TAK-831 50 μg (N=6) | [14C]TAK-831 500 mg (N=6)
Eye irritation (Eye disorders) | 0 | 0 | 1
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Generally, the PI may publish results of the study following the publication of results by the Sponsor.

DOCUMENTS (2):
  • Study Protocol (2019-10-29): https://cdn.clinicaltrials.gov/large-docs/72/NCT04234672/Prot_000.pdf
  • Statistical Analysis Plan (2020-04-16): https://cdn.clinicaltrials.gov/large-docs/72/NCT04234672/SAP_001.pdf